CLINICAL TRIAL: NCT05755464
Title: Validation of a Collaboration Evaluation Form for the Purposes of Dental and Orthodontic Treatment of the Patient With Down Syndrome
Brief Title: Evaluation of Patients With Down Syndrome Compliance to Dental Therapy
Status: Suspended | Type: Observational
Why Stopped: Reorganization of the clinic
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 1946
Record Dates: First submitted 2023-02-06; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Down Syndrome
Keywords: Down Syndrome; Dental disease; Compliance
MeSH Terms: conditions — Down Syndrome; Stomatognathic Diseases; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since subjects with Down Syndrome (DS) have different and variable levels of intellectual deficit, in approaching the patient with DS and before evaluating the different therapeutic strategies and carrying out a dental and orthodontic treatment, an initial analysis would be useful the patient's level of cooperation.

The hypothesis underlying the study is the possibility of predicting the degree of success of dental and orthodontic treatment in the patient with Down's Syndrome by completing an evaluation form by the clinician. The general objective of the study is to test the effectiveness of the module in assessing and quantifying the degree of patient collaboration.

This form is filled in entirely during the first visit and updated in subsequent sessions in conjunction with the different operational phases.

Based on the score obtained by the patient, the clinician can hypothesize the degree of cooperation during the operative sessions and compliance with the indications provided.

Therefore, the evaluation of the score obtained will guide the clinician in choosing the type of therapy that will have the least risk of failure because this will be chosen having evaluated not only the dental and/or orthodontic therapeutic needs, but also the real ability of the patient to collaborate.

DETAILED DESCRIPTION:
In the planning and management of dental and/or orthodontic treatments aimed at people with intellectual disabilities, the role of the clinician and his ability to empathize with the patient in order to obtain collaboration in treatment is fundamental. For these reasons it is necessary that, before planning the therapy, he can carry out a careful and complete evaluation of the behavioral profile that these subjects manifest.

Given the scarce presence in the literature of studies relating to an a priori evaluation of patient collaboration, this study aims to propose an objective and reproducible protocol to evaluate the patient's behavioral typology at the beginning of the treatment relationship, so as to improve the quality of the diagnosis and subsequent treatment of the patient by directing the clinician towards the most appropriate and effective treatment.

Down syndrome (DS), which our study deals with, is the result of trisomy of chromosome 21, and is considered the main genetic cause of mental disability. Trisomy of chromosome 21 affects both physical and cognitive development and results in a characteristic behavioral phenotype; however, the individuals concerned show a great variability of behavior in relation to the severity of the specific deficit, and this affects the chances of success of a dental treatment and, if necessary, the success and stability in the short and long term long-term orthodontic treatment.

In subjects with Down syndrome orofacial dyskinesia has a high prevalence and consists of a set of abnormal and involuntary movements of the facial muscles and/or masticatory muscles, which determine mandibular movements in protrusion and bruxism. Due to the marked orofacial hypotonia, the subject encounters considerable difficulties in sucking, swallowing, speaking and chewing from the first years of life. For this reason, an intervention aimed at solving the problems relating to swallowing, phonation, breathing and chewing is necessary, since these anomalies can preclude the possibility of a normal integration into the social context and relationship life by these subjects.

Furthermore, obstructive sleep apnea syndrome (OSAS) is significantly more prevalent among children with DS than in the general population, and a bidirectional and complex link between sleep disturbances and pediatric health has been demonstrated: sleep disturbances they have been associated with the development of obesity and cardiovascular abnormalities, epilepsy, autism spectrum disorders, attention deficit hyperactivity disorder (ADHD), mood and anxiety disorders, and a wide range of neurocognitive problems.

At the level of the oral cavity, a greater prevalence of oligodontia has been demonstrated in subjects with Down syndrome: the teeth that are most frequently missing are the third molars, followed by the second premolars and the incisors. Some patients may also have deciduous teeth even in adulthood. Individuals with Down syndrome also have microdontia affecting all teeth except the upper first molars and lower incisors. A higher prevalence of class III malocclusion can also be observed in these individuals compared to the general population; this could be attributed to altered skull-to-bone ratios, reduced size of the dental arches, and decreased jaw size in patients with Down syndrome. Another interesting fact is that these subjects show a higher incidence of fractures of the dental elements than the general population, mainly affecting the upper incisors, due to the greater frequency of severe maxillary overjet, class II-I division malocclusion, short or incompetent superior and a greater accident proneness.

At the craniofacial level in the subject with DS the height of the palate is significantly reduced and the presence of a "torus palatine" can easily be found which gives the palate a characteristic "W" shape; this is frequently associated with upper airway obstruction. The presence in such subjects of a high arched palate and the reduction of the nasal septum contribute to a considerable narrowing of the nasal antrum and therefore limit the development of the upper airways. Because of this, children with DS are forced to breathe through their mouths and maintain a low tongue posture and are therefore termed oral breathers. Therefore, the lack of ventilation of the upper airways does not cause the flattening action of the floor of the nasal cavities operated by the air flow. In oral respirator it is also important to evaluate the state of the adenoids, the presence of hypertrophic tonsils and any allergic diseases (allergic rhinitis, bronchial asthma). Furthermore, in a study by Oliveira et al. it was observed that at the oral level there was a direct correlation between the presence of airway infections in the 6 months prior to the trial and an increased risk of 2.47 of developing posterior crossbite.

Untreated oral respiratory subjects may develop a distinctive facial profile, with long narrow faces, narrow jaws, a high-arched palate with dental malocclusion, a gingival smile, and skeletal class III. For these reasons, an early and specific orthodontic treatment is essential: the expansion of the palate in fact determines an increase in the nasal volume and in the ability to implement nasal rather than oral breathing.

For these reasons, an adequate medical approach, combined with early dental intervention, can lead to a reduction in the prevalence of malocclusions in subjects with DS, with a consequent beneficial effect on the development of these subjects. In order to improve the oral health of these individuals, defined as "special needs patients", it is essential that the public health services that deal with oral health introduce intervention methods dedicated to the prevention and treatment of malocclusions. It is therefore essential to understand the panorama of the dental needs of people with disabilities in order to ensure treatments that can help this component of the population overcome difficulties and improve their growth opportunities and quality of life.

In these subjects it is possible to find deviations from the norm with regard to the size, shape or position of the maxilla and mandible. The types of malocclusion most commonly found in these subjects are dental crowding, open bite, mono- or bilateral crossbite and skeletal class III. Malocclusion in these subjects not only negatively affects functions such as chewing, language, sucking and swallowing, but also has important consequences on the psychological profile due to unacceptable dental aesthetics.

The implementation of orthodontic treatments in subjects with DS has the objective of restoring normal masticatory function and of creating greater resistance to the disease and an overall improvement of the personal appearance, which contributes positively to the physical and mental well-being of the subject. In fact, analyzing the picture in relation to the aesthetic aspect, it can be observed how the presence of bad breath, dental malposition, trauma, gum bleeding, open mouth posture and excessive salivation can lead to feelings of compassion or repugnance and discrimination from others individuals, thus accentuating a tendency to isolate these subjects from the life of society.

The patient with Down syndrome represents an ideal candidate to carry out a study aimed at evaluating the collaboration in dental and orthodontic treatments, since he presents a series of peculiar orthodontic anomalies, such as 3rd class malocclusion, open bite, cross bite and agenesis; it has also been observed that subjects with DS show a very different degree of collaboration based on the severity of the developmental and behavioral deficits. Consequently, some of them will show a more positive and favorable attitude towards dental care, while others will be treatable with more difficulty or treatable exclusively in partial or total sedation. For these reasons, although the need for orthodontic treatment is often present, this is not always feasible until all the treatment objectives have been achieved: in fact, often, due to the poor collaboration of patients with Down syndrome, partial objectives are established and /or minimally invasive orthodontic means are used with limited results.

ELIGIBILITY:
Inclusion Criteria:

* Down Syndrome
* Need of Dental treatment
* malocclusion

Exclusion Criteria:

* other existing pathologies

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study is expected to evaluate 100 Italian patients aged between 9 and 16 years with DS, who require an evaluation of dental malocclusion and orthodontic correction.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of a module designed to evaluate the level of collaboration of the dental patient with DS. | 3 years
  The aspects that, during the procedures, are indicative of the collaboration, translated into numerical values are counted.

CONTACTS AND LOCATIONS:
Locations (1):
- Università Cattolica del Sacro Cuore, Rome, Italy

IPD SHARING:
Plan to Share IPD: No